CLINICAL TRIAL: NCT06540365
Title: Feasibility and Effectiveness of the Pathways and Resources for Engagement and Participation Protocol Among Youth and Young Adults With Duchenne and Becker Muscle Dystrophies- A Pilot Study
Brief Title: Applying the Pathways and Resources for Engagement and Participation Protocol Among People With Muscles Dystrophies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Michal Waisman Nitzan, Faculty member, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBMD PREP Intervention
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Health Resources

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-Based activity program (Experimental)
  Interventions: Behavioral: Pathways and Resources for Engagement and Participation (PREP)

INTERVENTIONS:
Behavioral: Pathways and Resources for Engagement and Participation (PREP) — Each participant will work individually with an occupational therapist (OT) to pursue one leisure-oriented, community-based activity chosen by the young person. The participant will choose the community program using the PREP 5 steps (Make goals; Map out a plan; Make it happen; Measure the process and outcomes; Move forward). The OT will then search for the appropriate program, identify and remove potential environmental barriers to participation in that activity (e.g., accessibility, equipment), and educate program instructors regarding the person's specific needs. This process will include an expected 8 sessions lasting 12 to 18 weeks (depending on the assigned baseline length).

SUMMARY:
Taking part in community activities is essential for health and well-being. Yet, it is highly restricted for young people with Duchenne and Becker Muscular Dystrophies (DBMD), especially as they grow into adulthood. The Participation Pathways and Resources for Engagement and Participation (PREP) intervention is designed to help remove barriers in the environment.

This study aims to see if the PREP intervention is useful and practical for youth and young adults with DBMD. The main question is: How useful is the PREP intervention for improving participation in community-based activities chosen by the participants? Participants will start the study at different times (4, 5, or 6 weeks) and work one-on-one with an occupational therapist on a leisure activity of their choice. They will have eight sessions over 12 to 18 weeks to work on this activity.

They will use the Canadian Occupational Performance Measure (COPM) every week to track their performance and satisfaction with the chosen activity before, during, and after the intervention. The findings of this study can guide clinicians, families, and policymakers to select effective approaches that promote the participation of youth and young adults with DBMD in 'real world' activities they choose. It can also increase motivation and compliance and reduce the burden on the healthcare system, families, and people with DBMD themselves.

DETAILED DESCRIPTION:
Duchenne-Becker muscular dystrophy (DBMD) is an X-linked recessive disorder affecting 1 in 5,000 to 1 in 6,000 live male births, resulting in difficulties with movement and multi-system implications. The affected physical abilities deteriorate as the child grows up. In many cases, the use of a wheelchair is required at around 10 to 12 years of age, followed by a deterioration of strength in the upper limbs and cardiac complications. During the last decade, the average life expectancy of people with DBMD has risen to their forties. As participation in self-chosen meaningful activities within the community and society is essential to health and well-being, there is a need to address new opportunities for people with DBMD to participate in an independent and fulfilling life. Specifically, this pilot study will examine the effectiveness of the PREP intervention protocol among youth and young adults with DBMD.

A single-subject experimental design with multiple baselines across participants will be used to study the relative effect of the intervention. The intervention will be implemented for 6 participants with DBMD aged 14 to 30 and will be introduced at varying times. Every two participants will be randomly assigned to 3 baseline lengths (4, 5, 6 weeks). By varying the length of the baseline phase across participants, extraneous variables such as maturation and carry-over effects are controlled for. Each participant will work individually with an occupational therapist on one participation goal related to leisure-oriented community-based activity chosen by the young person, on expected eight sessions throughout 12 to 18 weeks (depending on the assigned baseline length). The participants will complete the Canadian Occupational Performance Measure weekly through all study phases (baseline + intervention).

For each participation goal, a series of data points representing the level of goal performance and satisfaction generated from the COPM will be plotted and analyzed to detect change. Visual analysis will be used to identify and compare patterns of change (e.g., level, variability, and trend) between the baseline and intervention phases. A statistical analysis will be used to complement visual interpretation. Specifically, an acceleration line will detect a trend and slope change across intervention phases. This method calculates the proportion of data points falling above and below the line. If 50% are above the line and 50% below the line, this result indicates no treatment effect, whereas significantly more observations falling above the line indicate a change in goal performance.

The research team, comprised of researchers in the field of complex disabilities and transition-aged youth and young adults, has partnered with the Little Steps Association for Children with Duchenne and Becker Muscular Dystrophy and is well-positioned to accomplish the study objectives.

This study will draw initial conclusions to support effective approaches that promote the participation of youth and young adults with DBMD in 'real world' activities they choose. Findings can also suggest implications such approaches can have on increasing motivation and compliance of people with DBMD to intervention and reducing the burden on the healthcare system, families, and people with DBMD themselves.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with DBMD
* aged 14-30 years
* from any sector of Israeli society.

Exclusion Criteria:

* have previously received the PREP intervention

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Up to 18 weeks (once a week, during base-line and intervention phase)
  A gold-standard 10-point scale that measures activity performance and satisfaction. The score ranges from 1 (unable to perform) to 10 (performs extremely well)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Waisman-Nitzan, Dr, Principal Investigator — University of Haifa